CLINICAL TRIAL: NCT00926835
Title: A Study to Investigate the Effect of Antidepressants on the Treatment for Korean Major Depressive Disorder (MDD) Patients
Brief Title: Effect of Antidepressants on the Treatment for Korean Major Depressive Disorder Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to patient recruitment difficulties
Sponsor: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Jun Tae-Youn, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIHWAF-CRCD-K-01
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Paroxetine; Escitalopram; Venlafaxine Hydrochloride; Bupropion; Lamotrigine; Mirtazapine; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Paroxetine (Experimental): Paroxetine monotherapy
  Interventions: Drug: paroxetine
- Escitalopram (Active Comparator): Escitalopram monotherapy
  Interventions: Drug: Escitalopram
- Venlafaxine (Active Comparator): Venlafaxine monotherapy
  Interventions: Drug: Venlafaxine XR
- Paroxetine+Bupropion (Active Comparator)
  Interventions: Drug: Paroxetine+Bupropion
- Paroxetine+Lamotrigine (Active Comparator)
  Interventions: Drug: Paroxetine+Lamotrigine
- Paroxetine+Lithium (Active Comparator)
  Interventions: Drug: Paroxetine+Lithium
- escitalopram+mirtazapine (Active Comparator)
  Interventions: Drug: Escitalopram+Mirtazapine
- Escitalopram+Aripiprazole (Active Comparator)
  Interventions: Drug: Escitalopram+Aripiprazole
- Paroxetine + Venlafaxine (Active Comparator)
  Interventions: Drug: Paroxetine + Venlafaxine XR

INTERVENTIONS:
Drug: paroxetine — 6 weeks, 20-50mg/day
  Other Names: Seroxat
  Arms: Paroxetine
Drug: Escitalopram — 10-20mg/day for 6 weeks
  Other Names: lexapro
  Arms: Escitalopram
Drug: Venlafaxine XR — Venlafaxine 75-225mg/day for 6 weeks
  Other Names: Efexor XR
  Arms: Venlafaxine
Drug: Paroxetine+Bupropion — paroxetine 20-50mg/day + bupropion 150-400mg/day for 6 weeks
  Other Names: Seroxat, wellbutrin
  Arms: Paroxetine+Bupropion
Drug: Paroxetine+Lamotrigine — Paroxetine 20-50mg/day + lamotrigine 100-400mg/day for 6 weeks
  Other Names: seroxat, lamictal
  Arms: Paroxetine+Lamotrigine
Drug: Paroxetine+Lithium — Paroxetine 20-50mg/day + lithium 0.5-1.2 mEq/L
  Other Names: seroxat, lithan
  Arms: Paroxetine+Lithium
Drug: Escitalopram+Mirtazapine — escitalopram 10-20mg/day + mirtazapine 15-45mg/day for 6 weeks
  Other Names: lexapro, remeron
  Arms: escitalopram+mirtazapine
Drug: Escitalopram+Aripiprazole — escitalopram 10-20mg/day + aripiprazole 5-15mg/day for 6 weeks
  Other Names: lexapro, abilify
  Arms: Escitalopram+Aripiprazole
Drug: Paroxetine + Venlafaxine XR — Paroxetine 20-50mg/day + Venlafaxine 75-225mg/day for 6 weeks
  Other Names: seroxat, efexor XR
  Arms: Paroxetine + Venlafaxine

SUMMARY:
The primary purpose of this study is to investigate the effectiveness of antidepressants on the treatments for non-psychotic major depressive disorder (MDD) in Korea. The study divides MDD patients into 3 level groups according to their past histories to treatments and compares the effectiveness of various treatment regimens at each level.

The treatment level groups are: 1) patients who have never been treated with appropriate medications for their current depressive symptoms before, 2) who received an appropriate SSRI (Selective Serotonin Reuptake Inhibitor) once but did not respond to it, 3) who received two types of SSRI antidepressant treatments without much effects in reducing their depressive symptoms.

The first level group will be treated with a single SSRI antidepressant treatment. The second and third level groups, who received SSRI treatment before, will be treated with alternative SSRI antidepressants (switching), combined multiple SSRI treatments (antidepressant combination), or SSRI treatments combined with mood stabilizer or anti-psychotics (augmentation). This study does not use placebos. Patients will visit 5 times for 6 weeks at each level for treatments. Patients will be evaluated for the severity of depressive symptoms, functional level, and side effects at each visit. Afterwards, the investigations will combine to monitor the patients depressive symptoms in every 3 months for the next 24 months. 18 nationwide university hospitals will participate in this study. This multi-site, prospective, and naturalistic study for patients with depression in Korea is a main project of 'Clinical Research Center for Depression' funded by the Ministry for Health, Welfare, and Family Affairs (MIHWAF) in Korea for a highly-qualified research achievement.

DETAILED DESCRIPTION:
Patients will be classified into 3 levels by their past therapeutic histories:

Level 1: Patients who do not receive an appropriate treatment for their current major depressive episode.

Level 2: Patients who never showed a satisfactory response to an adequate dosage of Paroxetine during a sufficient period of their current major depressive episode.

Level 3: Patients without a satisfactory response to two or more antidepressants including one of Paroxetine or Escitalopram for a sufficient period.

A satisfactory response means baseline HAM-D17 score was reduced over 50% or HAM-D17 score 10 or below and a sufficient period means 6 weeks.

Patients will be randomly assigned to the following treatment groups. Patients in level 1 will be randomly assigned to treatment groups among Paroxetine monotherapy, Escitalopram monotherapy, or Venlafaxine monotherapy.

Patients in level 2 will be enrolled who were medicated Paroxetine monotherapy in level 1 and assigned to one of the following 4 groups; Escitalopram monotherapy, Venlafaxine monotherapy, Paroxetine combined with Venlafaxine, or Paroxetine augmented with Lithium.

Patients in level 3 will be randomly assigned to one of the following 4 groups: 1) Either Paroxetine combined with Lamotrigine or Paroxetine combined with Bupropion if they resist two antidepressants including Paroxetine. 2) Either Escitalopram combined with Mirtazapine or Escitalopram combined with Aripiprazole if they resist two antidepressants including Escitalopram. 3) Patients who does not respond to both Paroxetine and Escitalopram will be randomly assigned to either 1) or 2).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-psychotic Major depressive disorder
* HAMD-17 score 14 or greater
* Age of 18 or greater and 65 or less

Exclusion Criteria:

* patients with current or past history of diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or psychotic disorder NOS
* patients with current psychotic features, eating disorders or obsessive-compulsive disorder
* patients with neurological disorder
* patients with medical condition that could interfere with everyday life activities
* pregnant or lactating women,
* patients with current other DSM-IV TR Axis I diagnosis other than MDD which needs inpatient care
* patients who treated with ECT for current depressive episode
* insufficient information of past treatment for current depressive episode
* patients who posed a serious suicidal risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Youn Jun, MD, PhD, Study Chair — Clinical research center for depression
Locations (1):
- Clinical research center for depression, Seoul, Seoul, South Korea